CLINICAL TRIAL: NCT04410484
Title: PREPARE-IBD: Physician Responses to Disease Flares and Patient Adaptation in Relation to Events in Inflammatory Bowel Disease During COVID-19 Pandemic
Acronym: PREPARE IBD
Status: Completed | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 284920
Record Dates: First submitted 2020-05-29; First posted 2020-06-01 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Inflammatory Bowel Diseases; Coronavirus Infection
MeSH Terms: conditions — Inflammatory Bowel Diseases; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1: Admitted patients with IBD (with IBD OR due to COVID) whether tested or not tested for COVID between 1st March and 30th June 2020
- 2: Patients with IBD self-isolating with suggestive COVID19 symptoms (Fever or persistent Cough) or tested positive for COVID19 during same period
- 3: Patients with active IBD identified during the same study period. (definition: increased symptoms suggestive of flare, raised calprotectin, raised CRP, endoscopy or imaging during the previous 6 weeks showing active disease and contacted/reviewed during the study period , admission with IBD ( These will be identified through your helpline/ virtual clinics/Hot clinics/flare lines
- Control Group: Consecutive patients with active IBD between 1st March 2019-30th June 2019

SUMMARY:
To find out what adaptations have been made by Inflammatory bowel disease physicians and patients in relation to therapies in flaring IBD patients during severe acute respiratory syndrome 2-COV and what the impact of these is on IBD patients with no symptomatic COVID-19 and in suspected/confirmed COVID-19. Also whether there any IBD related factors impacting the outcome of patients with COVID-19 symptoms or COVID-19 disease

DETAILED DESCRIPTION:
An observational, retrospective, case-controlled study to determine the status of IBD during development of COVID-19 symptoms/positive COVID-19. The aim is to describe the adaptations in therapies for active IBD during SARS COV 2 in patients with active IBD and positive or negative COVID-19 symptoms. It will evaluate IBD outcomes following development of COVID-19 symptoms / positive COVID-19 and determine any predictors of outcomes in IBD patients with COVID-19 symptoms / positive COVID-19 as well as determine the impact on IBD outcomes resulting from adaptations to treatments during COVID-19

ELIGIBILITY:
Inclusion Criteria:

* Patients with IBD +/- flare +/- COVID 19 positivity

Exclusion Criteria:

* Patients below 16
* Patient with inactive IBD

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: About 1 in 100- to 1 in 200 patients have IBD and up to 550,000 patients are estimated in the UK.
Sampling Method: Probability Sample
Enrollment: 3728 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Flare of IBD needing change in therapy or surgery | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Sebastian, Principal Investigator — Hull and East Yorkshire NHS Trust
Locations (1):
- Gastroenterology, Hull Royal Infirmary, Hull University Teaaching Hospitals NHS Trust, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Resulting publication — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9383326/